CLINICAL TRIAL: NCT03770416
Title: Nivolumab and Ibrutinib for Relapsed or Refractory Central Nervous System Lymphoma
Brief Title: Nivolumab and Ibrutinib in Treating Patients With Relapsed or Refractory Central Nervous System Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0510; NCI-2018-02181 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0510 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-12-04; First posted 2018-12-10 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Central Nervous System B-Cell Non-Hodgkin Lymphoma; Recurrent Central Nervous System Lymphoma; Refractory Central Nervous System Lymphoma
MeSH Terms: interventions — ibrutinib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A (Experimental): Patients receive ibrutinib PO daily on days 1-28. Beginning course 1, patients also receive nivolumab IV over 1 hour on days 1 and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve at least a partial response after 6 courses may continue therapy for up to 2 years.
  Interventions: Drug: Ibrutinib; Biological: Nivolumab
- Cohort B (Experimental): Patients receive ibrutinib PO daily on days 1-28 and nivolumab IV over 1 hour on days 1 and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve at least a partial response after 6 courses may continue therapy for up to 2 years.
  Interventions: Drug: Ibrutinib; Biological: Nivolumab

INTERVENTIONS:
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo

SUMMARY:
This phase II trial studies the side effects and how well nivolumab and ibrutinib works in treating patients with central nervous system lymphoma that has come back or does not respond to treatment. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Ibrutinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving nivolumab and ibrutinib may work better in treating patients with central nervous system lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the overall response rate of nivolumab and ibrutinib in central nervous system (CNS) lymphoma.

SECONDARY OBJECTIVES:

I. Determine the overall response rate of 4 weeks of ibrutinib single agent in CNS lymphoma.

II. Determine the complete response rate of nivolumab and ibrutinib in CNS lymphoma.

III. Determine the 1-year progression free and overall survival outcomes in CNS lymphoma.

IV. Safety and toxicity of nivolumab and ibrutinib.

EXPLORATORY OBJECTIVES:

I. Assess activation of T cells in peripheral blood and cerebrospinal fluid. II. Assess the cytokine profile from microglial cells in cerebrospinal fluid. III. Correlate features of peripheral blood T cell activation with toxicities. IV. Correlate features of peripheral blood T cell activation with response and progression free survival (PFS).

V. Correlate baseline tumor characteristics with response and PFS. VI. Evaluate the ability of minimal residual disease testing to monitor response and differentiate from pseudo progression.

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT A: Patients receive ibrutinib orally (PO) daily on days 1-28. Beginning course 1, patients also receive nivolumab intravenously (IV) over 1 hour on days 1 and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

COHORT B: Patients receive ibrutinib PO daily on days 1-28 and nivolumab IV over 1 hour on days 1 and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients who achieve at least a partial response after 6 courses may continue therapy for up to 2 years.

After completion of study treatment, patients are followed up within 3-4 weeks and then every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed refractory central nervous system lymphoma, pathology confirmed B cell lymphoma either by biopsy or by CSF review. Patient must previously have had at least one line of systemic therapy for CNS lymphoma.
2. Age 18 years or older
3. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤2
4. Patients must have adequate renal and hepatic function

   * Total bilirubin ≤1.5 x upper limit of normal (ULN). For patients with Gilbert's disease, total bilirubin up to ≤3 x ULN is allowed provided normal direct bilirubin.
   * Serum creatinine ≤1.5 x ULN
   * ALT and AST ≤3 x ULN
5. Females of childbearing potential must have a negative serum or urine beta human chorionic gonadotrophin (β-hCG) pregnancy test result within 24 hours prior to the first dose of treatment and must agree to use a highly effective contraception method during the study and for 23 weeks following the last dose of the study drugs. Females of non- childbearing potential are those who are postmenopausal greater than 1 year or who have had a bilateral tubal ligation or hysterectomy. Males who have partners of childbearing potential must agree to use an effective contraceptive method during the study and for 31 weeks following the last dose of study drugs. Men must agree not to donate sperm during and for 3 months after the last dose of study drug. Women who are pregnant or breastfeeding are ineligible for this study.
6. Patients or their legally authorized representative must provide written informed consent.
7. Hematology values must be within the following limits:

   1. Absolute neutrophil count (ANC) 1000/mm3 independent of growth factor support
   2. Platelets 100,000/mm3 or 50,000/mm3 if bone marrow involvement independent of transfusion support in either situation
8. Creatinine clearance (CrCl) > 30 ml/min

Exclusion Criteria:

1. History of another primary invasive malignancy that has not been definitively treated or in remission for at least 2 years. Patients with non-melanoma skin cancers or with carcinomas in situ are eligible regardless of the time from diagnosis (including concomitant diagnoses). If patients have another malignancy that was treated within the last 2 years, such patients may be enrolled if the likelihood of requiring systemic therapy for this other malignancy within 2 years is less than 10%, as determined by an expert in that particular malignancy at MD Anderson Cancer Center and after consultation with the Principal Investigator
2. Any major surgery or wound that has not healed, radiotherapy, cytotoxic chemotherapy, biologic therapy, immunotherapy, immunomodulatory drugs, experimental therapy within 4 weeks prior to the first dose of the study drugs.
3. Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification.
4. History of stroke or cerebral hemorrhage within 6 months of enrollment.
5. Patients who have uncontrolled hypertension (defined as sustained systolic blood pressure ≥ 160 mmHg or diastolic ≥ 100 mmHg)
6. Prior history of BTK inhibitor or PD1 inhibitor prior to start of trial.
7. Active, uncontrolled autoimmune hemolytic anemia or immune thrombocytopenia requiring steroid therapy.
8. Patients with autoimmune diseases are excluded: Patients with a history of Inflammatory Bowel Disease (including Crohn's disease and ulcerative colitis) are excluded from this study as are patients with a history of autoimmune disease (e.g., rheumatoid arthritis, systemic progressive sclerosis, systemic lupus erythematosus, Wegener's granulomatosis).
9. Patients with previous allogeneic stem cell transplant (SCT) within 6 months or with active acute or chronic graft-versus host disease are excluded. Patients must be off immunosuppression for GVHD for at least 30 days before cycle 1 day 1.
10. Patients with organ allografts (such as renal transplant) are excluded.
11. History of biopsy proven interstitial lung disease or pneumonitis which has impacted PFT in a clinically significant manner.
12. Patients who are on high dose steroids (>10mg daily of prednisone or equivalent) or immune suppression medications. Note: Patients on high-dose steroids (doses >10mg/day of prednisone or equivalent) or immune suppression medications are eligible provided these drugs are discontinued at least 3 days prior to starting on the study drugs.
13. Patients with uncontrolled active infection (viral, bacterial, and fungal) are not eligible.
14. Active current hepatitis B or C infection/reactivation as measured by DNA/RNA quantification, or known seropositivity for HIV.
15. Patient is pregnant or breast-feeding.
16. Malabsorption syndrome or other condition that precludes enteral route of administration.
17. Concomitant use of warfarin or other Vitamin K antagonists.
18. Requires chronic treatment with a strong cytochrome P450 (CYP) 3A inhibitor (see Appendix 3).
19. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and/or would make the patient inappropriate for enrollment into this study.
20. Vaccinated with live, attenuated vaccines within 4 weeks of enrollment.
21. Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to 2 years
  The overall response rate and its 95% confidence interval will be estimated. Fisher's exact test will be used to evaluate the association between response and other categorical patient variables.

SECONDARY OUTCOMES:
ORR | At 4 weeks of ibrutinib single agent
  The overall response rate and its 95% confidence interval will be estimated. Fisher's exact test will be used to evaluate the association between response and other categorical patient variables.
Progression free survival (PFS) | From study entry to objective disease progression or death from any cause, assessed at 1 year
  Will be estimated using the method of Kaplan and Meier.
Overall survival | From study entry to death, assessed at 1 year
  Will be estimated using the method of Kaplan and Meier.
Incidence of adverse events (AEs) | Baseline up to 30 days after the last dose of study drug
  AE data will be summarized by frequency tables for all patients. For the toxicity endpoint, per-treated analysis will be performed to include any patient who received the treatment regardless of the eligibility nor the duration or dose of the treatment received.

OTHER OUTCOMES:
T cells activation in peripheral blood and cerebrospinal fluid | Baseline up to 2 years
  Descriptive statistics including plots, mean, median and standard deviations will be used to summarize data. T-test and analysis of variance (ANOVA) will be used to compare outcome measures across patient characteristics. Dunnett's and Tukey's test that properly adjust for multiplicity in multiple tests will be implemented. Pair-wise comparisons will be performed using pre- and post-therapy samples from each patient. The chi-square (c2) test or Fisher's exact test will be used to test the association between two categorical variables such as disease state and performance status. Both univariate and multivariate logistic regressions will be performed to model prognostic factors.
Cytokine profile from microglial cells in cerebrospinal fluid | Baseline up to 2 years
  Descriptive statistics including plots, mean, median and standard deviations will be used to summarize data. T-test and ANOVA will be used to compare outcome measures across patient characteristics. Dunnett's and Tukey's test that properly adjust for multiplicity in multiple tests will be implemented. Pair-wise comparisons will be performed using pre- and post-therapy samples from each patient. The chi-square (c2) test or Fisher's exact test will be used to test the association between two categorical variables such as disease state and performance status. Both univariate and multivariate logistic regressions will be performed to model prognostic factors.
Tumor characteristics | Baseline up to 2 years
  Correlation baseline tumor characteristics with response and PFS will be calculated. Pair-wise comparisons will be performed using pre- and post-therapy samples from each patient. The chi-square (c2) test or Fisher's exact test will be used to test the association between two categorical variables such as disease state and performance status.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Westin, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Chihara D, Steiner RE, Nair R, Feng L, Ahmed S, Strati P, Malpica L, Griffith DP, Mathew SA, Montinez W, Masand G, Samaniego F, Rodriguez MA, Hagemeister FB, Fayad LE, Iyer SP, Nastoupil LJ, Neelapu SS, Flowers CR, Westin JR. Phase 2 trial of ibrutinib and nivolumab in patients with relapsed CNS lymphomas. Blood Adv. 2025 Apr 8;9(7):1485-1491. doi: 10.1182/bloodadvances.2024014635. PMID 39908461
- See also: M D Anderson Cancer Center — http://www.mdanderson.org